CLINICAL TRIAL: NCT05025683
Title: Analyzing Patient Flows at the Emergency Department by Data Analytics, Simulation, and Optimization
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Colin Graham, Professor, Chinese University of Hong Kong
Other Study IDs: CRE.2018.342
Record Dates: First submitted 2021-08-19; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Emergency Patients
Keywords: Emergency department; Simulation; Patient Flows
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this project, investigators apply operations research techniques, more specifically data analytics, system simulation, mathematical modelling, and optimization, for analyzing and improving operations in the Emergency Department at the Prince of Wales Hospital. The long term goals of this project are to demonstrate that integrated approach of data analytics and systems thinking is beneficial to health service planning and to extend present work to applications in other health-service systems.

DETAILED DESCRIPTION:
Design and subjects The current study requires time stamps for which patients start and end activities in the department. Personally identifiable information is not needed in this study. Investigators will collect the data from the computer system of the Department. The data will be used for data analysis and the development of simulation and optimization models. With current models, investigators investigate the effects of queueing policies, study workforce planning, and conduct a cost-effectiveness analysis for strategic planning.

Study instruments Data analytics tools and simulation and optimization softwares are needed in this research.

Interventions With simulation and optimization models, investigators examine the impacts of different operational strategies on the performance of the Emergency Department. The Computational experiments will not disturb the actual operations but will provide insights into the effectiveness of the various intervention policies.

Main Outcome Measures Investigators will derive insights from computational experiments and deliver useful recommendations for managing emergency department operations in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* All the patients attended to the Emergency Department of Prince of Wales Hospital in the period of July 2017 to June 2018 will be included in this study.

Exclusion Criteria:

* No patient will be excluded in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients attended to the Emergency Department of Prince of Wales Hospital in the period of July 2017 to June 2018 will be included in this study.
Sampling Method: Probability Sample
Enrollment: 23425 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Quantitative models | 12 months after recruitment
  Quantitative models, powered by domain knowledge of the Emergency Department (ED) system and ED operational data, will be developed to address three main operational problems in an ED: patient waiting time prediction, impacts of an adoption of a fast-track system, and patient scheduling

CONTACTS AND LOCATIONS:
Overall Officials: Colin A Graham, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, NT, Hong Kong